CLINICAL TRIAL: NCT04627506
Title: Role of Cerebral Oximetry in Reducing Postoperative End Organ Dysfunction/Failure After Complex Non-Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2019/00827
Record Dates: First submitted 2020-10-30; First posted 2020-11-13 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-09

CONDITIONS: Surgery
Keywords: Cerebral Desaturation

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, controlled clinical trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects will be randomly allocated to either interventional or control group according to a computer generated randomization code in predetermined size blocks.
  Bilateral NIRS (Masimo, O3TM Regional Oximetry) will be used to measure rSO2 intraoperatively. The NIRS screen will be concealed in the control group to ensure blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Bilateral NIRS will be used to measure rSO2 intraoperatively.
  In the control group, the cerebral oximetry monitor screen will be concealed, however, the recording will be continuous after verification of the signal strength and baseline value by an independent observer trained in cerebral oximetry application and unaware of the study design.
  Standardized anesthesia and surgical management will be conducted according to routine institutional practice.
- Study Group (Experimental): Bilateral NIRS will be used to measure rSO2 intraoperatively.
  In the interventional group, an alarm threshold at 90% of the baseline rSO2 value will be established. Based on predetermined algorithm the rSO2 will be maintained at or above 90% of the baseline measurements. The intervention will be commenced within 15 seconds of the reduction in rSO2 value.
  Interventions: Device: Bilateral NIRS (Masimo, O3TM Regional Oximetry)

INTERVENTIONS:
Device: Bilateral NIRS (Masimo, O3TM Regional Oximetry) — Bilateral NIRS will be used to measure rSO2 intraoperatively. The NIRS electrodes will be placed on fronto-temporal area and baseline values of rSO2 obtained according to manufacturer's guidelines in the operating room prior to induction of anesthesia. The NIRS screen will be concealed in the control group to ensure blinding.
  Arms: Study Group

SUMMARY:
The number of elderly patients requiring general anesthesia for major surgical procedures is increasing dramatically. It is estimated that 20% of these patients will develop major complications after surgery. Monitoring brain oxygen saturation may be helpful in reducing the postoperative complication rates. A decrease in brain oxygen is a sign that all other vital organs such as kidneys, heart, liver, and intestines have reduced blood supply and are starved from oxygen. This happens in 1 out of 5 patients undergoing major complex surgeries. Brain oxygen saturation monitor at this time is not used routinely during surgery, primarily due to the added cost, as well as, insufficient evidence that restoring the brain oxygen saturation to baseline would result in better outcomes. Patients will be randomly assigned to either study or control groups. In the study group, a special algorithm will be used to restore brain oxygen saturation. In the control group, the brain oxygen saturation will be monitored continuously, but the monitor screen will be electronically blinded, and standard clinical care applied. The objective of this study is to see if restoring the brain oxygen saturation to baseline results in less complication rates after surgery.

The objective of this study is to reduce the incidence of postoperative morbidity due to end organ dysfunction after major non-cardiac surgery in elderly patients.

The primary aim is to determine if restoration of rSO2 to baseline levels results in reduced incidence of major organ morbidity and mortality (MOMM).

A secondary aim is to determine a cost-effectiveness of this monitoring modality.

DETAILED DESCRIPTION:
With the increase in life expectancy observed in the last decades, the number of aged patients requiring general anesthesia for major non-cardiac surgery, such as abdominal, pelvic, and thoracic surgeries has increased dramatically. This patient population is at increased risk of postoperative complications due to the presence of multiple comorbidities and reduced physiological reserve. One of the largest prospective studies of over 4000 patients aged 70 years and over undergoing major non-cardiac surgery identified that 68% of these patients had pre-existing comorbidities. Furthermore, the 30-day postoperative mortality was 5% and major postoperative complications were present in 20% of patients. The authors concluded that strategies are needed to reduce complications and mortality in older surgical patients. The primary goal of hemodynamic management during the surgical procedure is to ensure adequate perfusion and oxygen delivery to the vital organs. In the last decade, technological research has expanded the application of near infrared spectroscopy (NIRS) to allow continuous non-invasive monitoring of cerebral oxygen saturation, providing information on the real time status on the balance between brain oxygen supply and demand. Furthermore, NIRS provides extra assurance of the adequacy of global oxygen balance, particularly focusing on the venous side of the circulation. Moreover several studies have demonstrated that changes in cerebral tissue oxygenation may correlate with changes in cerebral blood flow when cerebral metabolic rate of oxygen and arterial blood oxygen content remain constant. With the current standards of monitoring that primarily focus on the left heart, i.e., oxygen supply, and not the imbalance between oxygen supply/demand, the vital organ ischemia may go unnoticed until functional organ damage becomes evident. Regional cerebral oxygen saturation (rSO2) provides a non-invasive alternative of adequacy of systemic oxygen balance that correlates well with a gold standard of mixed venous oxygen saturation. Cerebral desaturations have been reported in more than 20% of cases when monitoring regional cerebral oxygen saturation (rSO2) in elderly patients undergoing non-cardiac abdominal surgery. Low rSO2 values have been associated with postoperative cognitive dysfunction (POCD), perioperative stroke, increased incidence of major organ morbidity, and even 30-day and 1-year mortality after cardiac surgery. Furthermore, low preoperative rSO2 measurements have been associated with higher risk of postoperative delirium in both cardiac and non-cardiac surgical populations. The proposed trial will be the first large prospective randomized controlled clinical trial assessing the effectiveness of rSO2 restoration in reducing postoperative morbidity associated with end organ dysfunction after major non-cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 60 years old
* Undergoing elective major non-cardiac surgery with predicted surgery length of 3 hours
* Signed informed consent

Exclusion Criteria:

* Emergency surgeries
* Laparoscopic / robotic surgeries
* Pregnant women

Ages: 61 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-02-18 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
A composite outcome of major end organ dysfunction | Surgery through to 6 months postoperatively
  A composite outcome will be assessed as a dichotomous outcome. (YES or NO). All components of the composite outcome will be weighted equally. They will include the following outcomes: postoperative delirium assessed with Confusion Assessment Method (CAM), Stroke assessed clinically, Transient Ischemic Attacks assessed clinically, Myocardial infarction, Pulmonary Embolism, Renal failure, Pneumonia, Atrial fibrillation, bleeding, mechanical ventilation for ≥48 hours, Major wound disruption, Surgical site infection, Sepsis, Septic shock, Systemic inflammatory response syndrome, Vascular graft failure. Frailty scale & DASI questionnaires will be administered at screening visit. Postoperative quality of recovery score (QoR-15) with be performed at baseline, POD 1 & 5 (discharge if earlier)]. Disability Free Survival (DFS) at 6 months (WHODAS).

CONTACTS AND LOCATIONS:
Overall Officials: Lian Kah Ti, Principal Investigator — National University Health System
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Story DA, Leslie K, Myles PS, Fink M, Poustie SJ, Forbes A, Yap S, Beavis V, Kerridge R; REASON Investigators, Australian and New Zealand College of Anaesthetists Trials Group. Complications and mortality in older surgical patients in Australia and New Zealand (the REASON study): a multicentre, prospective, observational study. Anaesthesia. 2010 Oct;65(10):1022-30. doi: 10.1111/j.1365-2044.2010.06478.x. PMID 20731639
- [Background] Casati A, Spreafico E, Putzu M, Fanelli G. New technology for noninvasive brain monitoring: continuous cerebral oximetry. Minerva Anestesiol. 2006 Jul-Aug;72(7-8):605-25. English, Italian. PMID 16865080
- [Background] Scott JP, Hoffman GM. Near-infrared spectroscopy: exposing the dark (venous) side of the circulation. Paediatr Anaesth. 2014 Jan;24(1):74-88. doi: 10.1111/pan.12301. Epub 2013 Nov 23. PMID 24267637
- [Background] Meng L, Cannesson M, Alexander BS, Yu Z, Kain ZN, Cerussi AE, Tromberg BJ, Mantulin WW. Effect of phenylephrine and ephedrine bolus treatment on cerebral oxygenation in anaesthetized patients. Br J Anaesth. 2011 Aug;107(2):209-17. doi: 10.1093/bja/aer150. Epub 2011 Jun 3. PMID 21642644
- [Background] Paarmann H, Heringlake M, Heinze H, Hanke T, Sier H, Karsten J, Schon J. Non-invasive cerebral oxygenation reflects mixed venous oxygen saturation during the varying haemodynamic conditions in patients undergoing transapical transcatheter aortic valve implantation. Interact Cardiovasc Thorac Surg. 2012 Mar;14(3):268-72. doi: 10.1093/icvts/ivr102. Epub 2011 Dec 7. PMID 22159266
- [Background] Green DW. A retrospective study of changes in cerebral oxygenation using a cerebral oximeter in older patients undergoing prolonged major abdominal surgery. Eur J Anaesthesiol. 2007 Mar;24(3):230-4. doi: 10.1017/S0265021506001645. Epub 2006 Oct 23. PMID 17054814
- [Background] Yao FS, Tseng CC, Ho CY, Levin SK, Illner P. Cerebral oxygen desaturation is associated with early postoperative neuropsychological dysfunction in patients undergoing cardiac surgery. J Cardiothorac Vasc Anesth. 2004 Oct;18(5):552-8. doi: 10.1053/j.jvca.2004.07.007. PMID 15578464
- [Background] Slater JP, Guarino T, Stack J, Vinod K, Bustami RT, Brown JM 3rd, Rodriguez AL, Magovern CJ, Zaubler T, Freundlich K, Parr GV. Cerebral oxygen desaturation predicts cognitive decline and longer hospital stay after cardiac surgery. Ann Thorac Surg. 2009 Jan;87(1):36-44; discussion 44-5. doi: 10.1016/j.athoracsur.2008.08.070. PMID 19101265
- [Background] Goldman S, Sutter F, Ferdinand F, Trace C. Optimizing intraoperative cerebral oxygen delivery using noninvasive cerebral oximetry decreases the incidence of stroke for cardiac surgical patients. Heart Surg Forum. 2004;7(5):E376-81. doi: 10.1532/HSF98.20041062. PMID 15799908
- [Background] Murkin JM, Adams SJ, Novick RJ, Quantz M, Bainbridge D, Iglesias I, Cleland A, Schaefer B, Irwin B, Fox S. Monitoring brain oxygen saturation during coronary bypass surgery: a randomized, prospective study. Anesth Analg. 2007 Jan;104(1):51-8. doi: 10.1213/01.ane.0000246814.29362.f4. PMID 17179242
- [Background] Heringlake M, Garbers C, Kabler JH, Anderson I, Heinze H, Schon J, Berger KU, Dibbelt L, Sievers HH, Hanke T. Preoperative cerebral oxygen saturation and clinical outcomes in cardiac surgery. Anesthesiology. 2011 Jan;114(1):58-69. doi: 10.1097/ALN.0b013e3181fef34e. PMID 21178669
- [Background] Schoen J, Meyerrose J, Paarmann H, Heringlake M, Hueppe M, Berger KU. Preoperative regional cerebral oxygen saturation is a predictor of postoperative delirium in on-pump cardiac surgery patients: a prospective observational trial. Crit Care. 2011;15(5):R218. doi: 10.1186/cc10454. Epub 2011 Sep 19. PMID 21929765